CLINICAL TRIAL: NCT00617695
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, 2-way Crossover Study With Single-blind, Placebo-challenge Evaluating the Efficacy of Zolmitriptan (Zomig) Nasal Spray 5mg, in the Treatment of Acute Migraine Headache in Adolescents.
Brief Title: Efficacy of Zolmitriptan (Zomig) in the Treatment of Migraines in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D1221C00005
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2009-04

CONDITIONS: Migraine
Keywords: Zolmitriptan; ZOMIG; migraine; headache response; headache; headache pain
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — zolmitriptan

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zolmitriptan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolmitriptan — 5mg nasal spray
  Other Names: Zomig
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Zolmitriptan (Zomig) nasal spray, 5.0 mg, compared with placebo (inactive drug) for 2 migraine headaches over a 3-month period in adolescent patients (aged 12 to 17 years) with migraine headaches

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-17 years at the time of screening. Patients must not be enrolled if they will turn 18 years of age within 12 weeks after randomization.
* An established diagnosis of migraine for at least 1 year; a minimum of 2 migraines, considered to be moderately/severely disabling, per month on average during the school year
* A history of usual migraine duration of >2-hours untreated for the 3 month prior to screening

Exclusion Criteria:

* A history of basilar, ophthalmoplegic or hemiplegic migraine headache or any potentially serious neurological condition that is associated with headache or clinically significant abnormalities indicated from the medical history, physical exam etc
* Has used monoamine oxidase inhibitor-A (MAO-A), methysergide, methylergonovine or cimetidine in the 2 weeks before randomization.
* Evidence of ischemic heart disease, arrhythmia, accessory conduction pathway disorder as determined by central cardiologist using predetermined and agreed upon pediatric standards; Has uncontrolled hypertension

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 247 (Actual)
Dates: Start 2003-09; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Headache response and pain-free response to treatment | 15 minutes, 30 minutes, 45 minutes, 1.5 hours and 2 hours after randomized treatment

SECONDARY OUTCOMES:
Adverse Event reports | Four times within 12 weeks